CLINICAL TRIAL: NCT06194981
Title: Duration of Postoperative Adjuvant Chemotherapy (3-4 Months Versus 5-6 Months) for Gastric Cancer Patients at Pathological N3 Stage: a Retrospective Study
Brief Title: Duration of Adjuvant Chemotherapy for Gastric Cancer Patients at Pathological N3 Stage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Hongyu Zhang, Attending doctor, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: 2023-KY-1488
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Capecitabine; S 1 (combination)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 3-4 months CapOx/SOX: Adjuvant CapOx/SOX 3-4 months after curative surgery:
  CapOx: Oxaliplatin: 130 mg/m²/day (day 1) , Capecitabine: 1,000 mg/m², bid (day 1-14), q3W, total 3-4 months (4-6 cycles); SOX: Oxaliplatin: 130 mg/m2/day(day 1) , S-1: 40-60 mg, bid (day 1-14), q3W, total 3-4 months (4-6 cycles)
  Interventions: Drug: Oxaliplatin and capecitabine/ S-1 and capecitabine
- 5-6 months CapOx/SOX: Adjuvant CapOx/SOX 5-6 months after curative surgery:
  CapOx: Oxaliplatin: 130 mg/m²/day (day 1) , Capecitabine: 1,000 mg/m², bid (day 1-14), q3W, total 5-6 months (7-8 cycles); SOX: Oxaliplatin: 130 mg/m2/day(day 1) , S-1: 40-60 mg, bid (day 1-14), q3W, total 5-6 months (7-8 cycles)
  Interventions: Drug: Oxaliplatin and capecitabine/ S-1 and capecitabine

INTERVENTIONS:
Drug: Oxaliplatin and capecitabine/ S-1 and capecitabine — Drug: capecitabine: 1000 mg/m² bid, po, d1-14, oxaliplatin: 130mg/m², iv drip for 2h, d1; S-1: BSA<1.25m², 40mg bid, 1.25m²≤BSA≤1.5m², 50mg bid, BSA>1.5m², 60mg bid, po, d1-14, oxaliplatin: 130mg/m², iv drip for 2h, d1
  Other Names: Xeloda

SUMMARY:
The goal of this retrospective study is to compare the efficacy and safety of 3-4 months to 5-6 months of CapOx/SOX adjuvant chemotherapy in pathological N3 gastric cancer patients.

DETAILED DESCRIPTION:
Due to a heavy metastatic node burden, pathological stage N3 (pN3) gastric cancer (GC) patients have extremely poor prognoses. Except for surgical resection, postoperative adjuvant chemotherapy is the major treatment strategy to improve survival for these patients. Capecitabine plus oxaliplatin (CapOx) and S-1 plus oxaliplatin (SOX) were considered the effective treatment for stage II and III GC after D2 gastrectomy in the CLASSIC and RESOLVE trials. But N3b (positive lymph nodes ≥16) and T1-3N3 patients were omitted in these two trials, respectively. Moreover, only 66.5% of patients finished 6 months of chemotherapy in the CLASSIC trial, and in the RESOLVE trial, 17-19% of patients required dose reductions and about 19% of patients discontinued chemotherapy due to drug-related toxicity for 6 months of chemotherapy. Particularly, cumulative administration of oxaliplatin led to peripheral sensory neurotoxicity, which caused poor quality of life and treatment compliance. Recently, a prospective analysis of six randomized, phase 3 trials with 12834 participants (IDEA trail) for stage III colon cancer, demonstrated that 3 months of CapOx was as effective as 6 months with relatively lower recurrence risk, no significantly different overall survival, and fewer adverse effects. However, there were no relevant studies to explore the optimal duration of chemotherapy for pN3 GC patients.

This study aims to compare the efficacy and safety of 3-4 months to 5-6 months of CapOx/SOX adjuvant chemotherapy in pathological N3 gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old
2. Pathological stage N3 GC (≥7 positive lymph nodes) after curative surgery according to the AJCC TNM staging system, 8th edition
3. Histologically confirmed R0 resection, defined as no macroscopic or microscopic residual tumor
4. Postoperative chemotherapy with CapOX or SOX doublet regimen, initiating within 6 weeks after curative gastrectomy
5. No distant metastases or gastric stump cancer
6. No other malignant tumors

Exclusion Criteria:

1. Patients who had undergone neoadjuvant chemotherapy or radiotherapy
2. Patients who received capecitabine or S-1 alone or combined with biological therapy, radiation therapy, or Immunosuppressive therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastric cancer patients who underwent D2 or D2+ procedure and pathologically confirmed stage N3 (AJCC 8th edition)
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2024-03-28 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 3 years
  The overall survival (OS) will be calculated from the day of surgery to participant's death with any cause

SECONDARY OUTCOMES:
Disease Free Survival | 3 years
  The Disease Free Survival (DFS) will be calculated from the day of surgery to participant's recurrence or death with any cause
Adverse Events | 6 months
  Adverse Events of Chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Hongyu Zhang, M.D., Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Department of Gastrointestinal Surgery, the First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No
Research data can be available through contacting the PI

REFERENCES:
- [Background] Noh SH, Park SR, Yang HK, Chung HC, Chung IJ, Kim SW, Kim HH, Choi JH, Kim HK, Yu W, Lee JI, Shin DB, Ji J, Chen JS, Lim Y, Ha S, Bang YJ; CLASSIC trial investigators. Adjuvant capecitabine plus oxaliplatin for gastric cancer after D2 gastrectomy (CLASSIC): 5-year follow-up of an open-label, randomised phase 3 trial. Lancet Oncol. 2014 Nov;15(12):1389-96. doi: 10.1016/S1470-2045(14)70473-5. Epub 2014 Oct 15. PMID 25439693
- [Background] Zhang X, Liang H, Li Z, Xue Y, Wang Y, Zhou Z, Yu J, Bu Z, Chen L, Du Y, Wang X, Wu A, Li G, Su X, Xiao G, Cui M, Wu D, Chen L, Wu X, Zhou Y, Zhang L, Dang C, He Y, Zhang Z, Sun Y, Li Y, Chen H, Bai Y, Qi C, Yu P, Zhu G, Suo J, Jia B, Li L, Huang C, Li F, Ye Y, Xu H, Wang X, Yuan Y, E JY, Ying X, Yao C, Shen L, Ji J; RESOLVE study group. Perioperative or postoperative adjuvant oxaliplatin with S-1 versus adjuvant oxaliplatin with capecitabine in patients with locally advanced gastric or gastro-oesophageal junction adenocarcinoma undergoing D2 gastrectomy (RESOLVE): an open-label, superiority and non-inferiority, phase 3 randomised controlled trial. Lancet Oncol. 2021 Aug;22(8):1081-1092. doi: 10.1016/S1470-2045(21)00297-7. Epub 2021 Jul 9. PMID 34252374
- [Background] Grothey A, Sobrero AF, Shields AF, Yoshino T, Paul J, Taieb J, Souglakos J, Shi Q, Kerr R, Labianca R, Meyerhardt JA, Vernerey D, Yamanaka T, Boukovinas I, Meyers JP, Renfro LA, Niedzwiecki D, Watanabe T, Torri V, Saunders M, Sargent DJ, Andre T, Iveson T. Duration of Adjuvant Chemotherapy for Stage III Colon Cancer. N Engl J Med. 2018 Mar 29;378(13):1177-1188. doi: 10.1056/NEJMoa1713709. PMID 29590544
- [Background] Andre T, Meyerhardt J, Iveson T, Sobrero A, Yoshino T, Souglakos I, Grothey A, Niedzwiecki D, Saunders M, Labianca R, Yamanaka T, Boukovinas I, Vernerey D, Meyers J, Harkin A, Torri V, Oki E, Georgoulias V, Taieb J, Shields A, Shi Q. Effect of duration of adjuvant chemotherapy for patients with stage III colon cancer (IDEA collaboration): final results from a prospective, pooled analysis of six randomised, phase 3 trials. Lancet Oncol. 2020 Dec;21(12):1620-1629. doi: 10.1016/S1470-2045(20)30527-1. PMID 33271092